CLINICAL TRIAL: NCT02334384
Title: Safety and Tolerability Study of Antimicrobial TheraGauze for Skin Abscess
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Eastern Virginia Medical School (Other)
Collaborators: Solsys Medical LLC (Industry); United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Kenji Cunnion, Associate Professor, Eastern Virginia Medical School
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SS-ATG-001
Record Dates: First submitted 2015-01-05; First posted 2015-01-08 (Estimated); Results first posted 2018-08-29 (Actual); Last update posted 2018-10-04 (Actual); Status verified 2018-09

CONDITIONS: Furunculosis
MeSH Terms: conditions — Furunculosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Antimicrobial TheraGauze (Experimental): Antimicrobial TheraGauze (i.e. tobramycin impregnated TheraGauze) will be used as a wound packing after incision and drainage of skin abscess (i.e. furunculosis). Antimicrobial TheraGauze will be administered once.
  Interventions: Biological: Antimicrobial TheraGauze
- Standard of care - standard wound packing (No Intervention): In this control arm the subject will receive standard of care with standard wound packing. The ED physician will have the choice to use plain cotton wick or iodoform wick. Standard wound packing will be administered once.

INTERVENTIONS:
Biological: Antimicrobial TheraGauze — In the intervention arm: Antimicrobial TheraGauze, tobramycin impregnated TheraGauze, will be used to pack the wound cavity after incision and drainage of the skin abscess.
  In the comparator arm: Standard wound packing, plain cotton wick or iodoform gauze - at the discretion of the provider will be used to pack the wound cavity after incision and drainage of the skin abscess.
  Arms: Antimicrobial TheraGauze

SUMMARY:
The goal of this study is to demonstrate safety and tolerability of a novel antimicrobial wound dressing, Antimicrobial TheraGauze. The unique microvillous structure of TheraGauze is ideal for the development of an antimicrobial wound dressing. In vitro testing has demonstrated that tobramycin is an ideal compound for integration into TheraGauze providing excellent killing of MRSA and other organisms that commonly cause wound infections. Tobramycin is a non-absorbable aminoglycoside that will be contained solely to the wound bed preventing any potential for systemic toxicities. In vivo testing of tobramycin-impregnated TheraGauze used in mouse wound models has confirmed no systemic absorption of tobramycin as demonstrated by undetectable blood levels. TheraGauze has been commercially available for 10 years as a wound dressing. Tobramycin has been available for many years as a topical antibiotic as eyedrops and as an inhaled antibiotic for patients with cystic fibrosis, demonstrating excellent safety in both cases.

This Phase I trial will test Antimicrobial TheraGauze (ATG) as an antimicrobial wound packing for patients presenting to an Emergency Department with skin abscess (furunculosis). Subjects will either receive ATG or standard of care wound packing (cotton wick or iodoform wick). Subjects will return to the ED in 2 days for wound packing removal and reassessment of their wounds and symptomatology. A final followup will be performed by a physician and study coordinator in an outpatient setting on day 7.

DETAILED DESCRIPTION:
Primary Endpoint. The primary endpoint of the study is to evaluate the safety of and identify side effects of TheraGauze/tobramycin wound packing compared with standard of care management for cutaneous abscesses requiring incision and drainage.

Methods.

Design:

This is a proof-of-concept, prospective, randomized clinical trial for safety of TheraGauze-tobramycin in adult subjects who present to Emergency Department settings for care of skin abscess requiring incision and drainage. A control, standard of care, arm is included to provide some data with respect to the side effect profile of current furunculosis management for comparison.

Two arms are proposed for this study:

1. Incision + TheraGauze+tobramycin packing (no systemic antibiotics)
2. Incision + standard iodoform wick or plain cotton wick packing (± p.o. antibiotics)

Anti-microbial TheraGauze (saturated tobramycin solution at 3 mg/ml) will be packed into the drained wounds of the subjects in the study arm. The control arm will receive current standard of care wound packing with a choice of iodoform wick or plain cotton wick, based on the preference of the ED physician. After packing, the wound excess TheraGauze or wick will be cut away. The ED physicians have the option to prescribe an oral antibiotic or not, according to their preference. The following oral antibiotic choices are available for subjects in the control arm only:

* Bactrim (TMP/SMX)
* Vibramycin (doxycycline)
* Cleocin (clindamycin) Antibiotics will be purchased by subjects from their local pharmacy.

TheraGauze-tobramycin. We plan to use TheraGauze saturated with tobramycin at 3 mg/ml, the same dose used in the ophthalmic preparations (e.g., Tobrex) and much smaller concentration than the concentration in tobramycin bone cement (50 - 60 mg/ml). The decades of efficacy and safety with tobramycin eye drops justifies using the 3 mg/ml concentration. In vitro testing with TheraGauze/tobramycin (0.9 mg/ml), shows excellent broad-spectrum antibacterial activity against Gram-negative and Gram-positive bacterial pathogens including all clinical MRSA strains tested (Echague, Hair et al. 2010). We expect that >85% of the cutaneous abscesses (furuncles) will be infected with MRSA (Demos, McLeod et al. 2012). Additionally, tobramycin is a non-absorbable antibiotic and thus an excellent choice for achieving local antimicrobial activity with minimal risk of systemic side effects, which it is why it is the most common antibiotic bone cement.

The TheraGauze/tobramycin wound packing will be placed after the incision and drainage of the abscess and removed at the day 3 (± 1) follow up visit in the Emergency Department. TheraGauze/tobramycin will only be placed in the wound a single time.

Methods:

Study Population:

Subjects from the Hampton Roads region of southeastern Virginia will be recruited from the hospital emergency department site staffed by EVMS physicians at Sentara Norfolk General Hospital.

Study Size:

We anticipate screening 200 patients in order to enroll and randomize 100 subjects. Subjects will be randomized 2:1 to the TheraGauze+tobramycin or iodoform wick/ plain cotton wick, respectively. We anticipate 50 participants completing the study. The 50% retention rate is typical for emergency department populations.

Recruitment and Retention:

Subjects who present to Emergency Department setting for care of skin abscess requiring incision and drainage will be approached by on-site Study Coordinators for enrollment. Upon meeting eligibility criteria and willingness to participate, subjects/LARs will provide informed consent. A medical information release will be obtained from the subject so that outcomes data can be collected related to additional unscheduled visits or adverse events cared for outside the emergency department setting.

Women and minority participation:

Adults up to 65 years of age will be enrolled regardless of gender and minority status as long as they are fluent in English.

Randomization:

A study subject identification number will be assigned. Subjects will then be sequentially randomized to one of two treatment arms upon enrollment in a 2:1 ratio, using a prepared list.

Study Treatments

Visit 1 - Day 1:

* Informed consent will be obtained from subject.
* Review of Eligibility Criteria (Inclusion/Exclusion)
* Randomization to Treatment Arm
* Contact Information to include phone number(s), address, primary care provider will be collected.
* Treatment and discharge with instructions to return to the ED for revaluation per routine care. The typical schedule is for the patients to return to the ED 2 days after initial wound care (Study Day 3 ±1).

The following information will be collected and recorded on a hard copy Case Report Form at this visit.

* Subject ID number
* Demographics
* Medical history
* Characteristics of symptoms and history
* Abscess characteristics
* Procedure information
* Laboratory Assessments - Per standard clinical care the abscess contents will be sent for routine Gram stain, bacterial culture and susceptibility testing.
* If patient is to receive iodoform wick/plain cotton wick then the care provider will have the option of prescribing a p.o. antibiotic, as is frequently done in these clinical settings.

Visit 2 - Day 3 ±1: (ED)

Subjects' wound status will be evaluated. The following information will be collected:

* Questions about infection
* Bacterial burden in wound bed - Wound culture performed using quantitative methods for culturing wound base (Gardner, Frantz et al. 2006).
* Wound assessment
* Schedule follow-up visit in EVMS Clinical Research Unit in 5 ± 1 days

Visit 3 - Day 7 ± 1: (EVMS Clinical Research Unit):

Follow up on subjects' wound status. The following information will be collected:

* Questions about infection
* Wound assessment

Statistical Analysis Plan The data will be analyzed using SAS 9.4 software. All statistical tests will be two-sided with a significance level of 0.05. Patients who withdraw while on treatment will be included in the data analysis for each time point before withdrawal. Baseline and follow-up measurements of safety, tolerability, numbers of pathogenic bacteria, wound infection persistence or worsening, and gross effects on the rate of wound healing will be summarized using descriptive statistics such as mean, median, standard deviation, interquartile range, frequency, and percentage where appropriate. Normality assessments for the continuous variables will be completed using Shapiro-Wilk tests and stem-and-leaf plots.

Tests of equivalence between the TheraGauze + tobramycin and standard iodoform wick packing treatment groups will establish statistical significance if the two-sided 90% confidence interval for the difference falls within the limits (-δ, δ), where δ is the margin of clinically accepted difference. This analysis will determine whether the outcomes are equivalent between the TheraGauze+tobramycin and standard iodoform wick packing treatment groups.

Protection of Human Subjects:

This research involves the recruitment, enrollment and management of human subjects participating in research. Adults up to age 65 years at enrollment are being studied because adults commonly suffer skin abscesses. Study oversight by the investigators will assure compliance with all regulatory requirements for Institutional Review Board approval prior to the initiation of the study, and will obtain annual re-approval for study activities.

Potential risks and benefits to subjects and procedures to mitigate risks:

* Physical/Medical

  o Serious/Adverse Events - will be reported to EVMS IRB
* Confidentiality/PHI o All PHI will be maintained in an encrypted and password protected electronic file.

ASSESSMENT OF SAFETY Subjects must be seen by a physician or an appropriately trained healthcare professional at every study visit, and the evaluation must be documented.

Adverse Events. An AE is any untoward medical occurrence in a clinical investigation subject administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.

Causality Assessment. For all AEs, the PI will provide an assessment of causal relationship to the study drug. Causal relationship must be assessed by answering the following question: Is there a reasonable possibility the study drug caused the event?

Adverse Reaction. An AE assessed as likely having a causal relationship with the intervention (i.e., TheraGauze/tobramycin). Specifically focusing on local-toxicity adverse reactions, we will evaluate for increasing redness, increasing pain or a new rash at the site of the packed wound. Increasing pain or redness could be due to progression of the infection (cellulitis/abscess) or local toxicity or reaction to the tobramycin in the TheraGauze/tobramycin packing. This will be assessed by an Investigator. Increasing purulent drainage or the identification of new areas of fluctuance requiring an additional incision and drainage procedure will be assessed as progression of the infection rather than evidence of local toxicity or reaction to the tobramycin.

Severity Assessment. The PI must provide an assessment of the severity of each AE by recording a severity rating, which will be assessed as described below. Severity, which is a description of the intensity of manifestation of the AE, is distinct from seriousness, which implies a subject outcome or AE-required treatment measure associated with a threat to life or functionality.

Guidelines for Adverse Event Severity Assessments Mild. Minor awareness of signs or symptoms that are easily tolerated without specific medical intervention. Moderate. Discomfort that interferes with usual activities and may require minimal intervention.

Severe. Significant signs or symptoms that are incapacitating with an inability to work or perform routine activities and/or that require medical intervention.

Serious Adverse Events. An SAE is any untoward medical occurrence that at any dose: is life threatening, requires in-patient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity. Important medical events may be considered serious when, based on appropriate medical judgment, they may jeopardize the subject and may require medical or surgical intervention to prevent one of the outcomes listed in this definition. If a serious and unexpected AE occurs for which there is evidence suggesting a causal relationship between the drug and the event the event must be reported as a serious and unexpected suspected adverse reaction. SAE will be reported to the local IRB and the FDA within 5 calendar days.

Stopping Rules. Adverse reactions, including local-toxicity adverse reactions, or SAEs will lead to immediate return to the SNGH ED for assessment and removal of the TheraGauze/tobramycin wound packing. The investigator will assess the need for treatment of the adverse reaction or SAE and, if necessary, either treat or refer for treatment, as appropriate. The subject will continue with their scheduled follow up: Day 3 visit in the ED, Day 6 phone follow up, and Day7 visit in the EVMS Clinical Research Unit.

ELIGIBILITY:
Inclusion Criteria:

* Ages >18 to <65 years at time of enrollment
* Subject has skin abscess requiring incision and drainage
* Male or female
* Ability to read and understand the English language at a level sufficient to provide informed consent and comply with study requirements
* Subject is willing and able to comply with all study requirements

Exclusion Criteria:

* Systemic illness or deep-seated infection requiring inpatient admission
* Deep seated infection requiring referral to surgery
* Subject requires oral antibiotics for suspicion of systemic spread of infection (i.e. bacteremia)
* Allergy to any aminoglycoside antibiotic.
* An underlying medical condition that impairs normal immune function (e.g. AIDS, cancer, diabetes, lupus, rheumatoid arthritis, organ or marrow transplantation, ulcerative colitis, Crohn's disease)
* Subject is pregnant or breastfeeding and/or a woman of childbearing potential who is not surgically sterile, not at least 2 years postmenopausal, or does not practice contraception methods, unless sexually abstinent for the duration of the study.
* Subject has any medical or psychiatric condition, in the opinion of the investigator, could jeopardize the subject's health or compromise the subject's ability to participate in the study.
* Subject has prior treatment with antibiotics in the preceding 7 (seven) days.
* Currently taking or has taken oral or injection steroid medication (e.g. prednisone) in the past 30 (thirty) days
* Currently taking or has taken immune suppressing medications (e.g. methotrexate, Prograf, CellCept, Rapamune) in the past 30 (thirty) days
* Currently taking or has taken medications to treat cancer in the past 30 (thirty) days
* Subject is currently participating or has participated within the last two months in any study of an investigational drug or device.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2017-08-01 (Actual); Study Completion 2017-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenji M Cunnion, M.D., M.P.H., Principal Investigator — Eastern Virginia Medical School
Locations (1):
- Sentara Norfolk General Hospital, Norfolk, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Antimicrobial TheraGauze: Antimicrobial TheraGauze (i.e. tobramycin impregnated TheraGauze) will be used as a wound packing after incision and drainage of skin abscess (i.e. furunculosis). Antimicrobial TheraGauze will be administered once.
  Antimicrobial TheraGauze: In the intervention arm: Antimicrobial TheraGauze, tobramycin impregnated TheraGauze, will be used to pack the wound cavity after incision and drainage of the skin abscess.
  In the comparator arm: Standard wound packing, plain cotton wick or iodoform gauze - at the discretion of the provider will be used to pack the wound cavity after incision and drainage of the skin abscess.
- Standard Wound Packing: Standard wound packing will be used as the active comparator. The ED physician will have the choice to use plain cotton wick or iodoform wick. Standard wound packing will be administered once.
  Antimicrobial TheraGauze: In the intervention arm: Antimicrobial TheraGauze, tobramycin impregnated TheraGauze, will be used to pack the wound cavity after incision and drainage of the skin abscess.
  In the comparator arm: Standard wound packing, plain cotton wick or iodoform gauze - at the discretion of the provider will be used to pack the wound cavity after incision and drainage of the skin abscess.
Period: Overall Study
Arm/Group | Antimicrobial TheraGauze | Standard Wound Packing
Started | 4 | 2
Completed | 3 | 1
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Antimicrobial TheraGauze | Standard Wound Packing | Total
Number analyzed (Participants) | 4 | 2 | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 2 | 6
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Standard Deviation); unit: years] | 33 (12) | 33 (12) | 33 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 4
  Male | 1 | 1 | 2
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4 | 2 | 6
Diameter of induration [Mean (Full Range); unit: mm] | 32.5 [25 to 40] | 27.5 [25 to 30] | 30.8 [25 to 40]

OUTCOME MEASURES:

1. Primary Outcome: Number of Side-effects
Description: Evaluate for evidence of side-effects from Antimicrobial TheraGauze packing of skin abscess wounds compared with standard of care (i.e. cotton wick or iodoform wick). Tests for statistical significance will be made for multiple potential side-effects including: 1) erythema around the wound packing, 2) increased pain at the wound site, 3) increased tenderness around the wound 4) increased discharge from the wound, 4) new rash, and 5) fever.
Time Frame: 1 week
Measure: Count of Participants; unit: Participants
Arm/Group | Antimicrobial TheraGauze | Standard Wound Packing
Number analyzed (Participants) | 4 | 2
Participants | 4 | 2

ADVERSE EVENTS:
Time Frame: 1 week
Arm/Group | Antimicrobial TheraGauze | Standard Wound Packing
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/2
Other Adverse Events (participants affected / at risk) | 0/4 | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-30): https://cdn.clinicaltrials.gov/large-docs/84/NCT02334384/Prot_SAP_000.pdf